CLINICAL TRIAL: NCT04533360
Title: Seroprevalence of SARS CoV2 Antibodies Among Adults in Kingman AZ
Brief Title: Prevalence of COVID-19 Antibodies Kingman AZ
Status: Completed | Type: Observational
Sponsor: Kingman Regional Medical Center (Other)
Responsible Party: Principal Investigator, John Ashurst, Emergency Medicine Residency Program Director, Kingman Regional Medical Center
Other Study IDs: KRMC 0205
Record Dates: First submitted 2020-08-28; First posted 2020-08-31 (Actual); Last update posted 2022-03-31 (Actual); Status verified 2022-03

CONDITIONS: Covid19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Month
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Community Cohort 1: 1000 Participants from the community will be recruited to undergo serological testing for SARS-CoV2 Antibodies at time point 1.
  Interventions: Diagnostic Test: VITROS Anti-SARS-CoV-2 IgG test
- Community Cohort 2: 1000 Participants from the community will be recruited to undergo serological testing for SARS-CoV2 Antibodies at time point 2.
  Interventions: Diagnostic Test: VITROS Anti-SARS-CoV-2 IgG test
- Healthcare Provider Cohort 1: 500 hospital employees will be recruited to undergo serological testing for SARS-CoV2 Antibodies at time point 1.
  Interventions: Diagnostic Test: VITROS Anti-SARS-CoV-2 IgG test
- Healthcare Provider Cohort 2: 500 hospital employees will be recruited to undergo serological testing for SARS-CoV2 Antibodies at time point 2.
  Interventions: Diagnostic Test: VITROS Anti-SARS-CoV-2 IgG test

INTERVENTIONS:
Diagnostic Test: VITROS Anti-SARS-CoV-2 IgG test — The VITROS Anti-SARS-CoV-2 IgG test is a lateral flow immunoassay produced by Ortho-Clinical Diagnostics Inc.

SUMMARY:
The COVID-19 disease outbreak is a historic event that has challenged medical systems in the United States. Currently, most reports of confirmed cases rely on the testing of symptomatic patients. These estimates of confirmed cases miss individuals who have recovered from infection, with mild or no symptoms, and individuals with symptoms who have not been tested due to the limited availability of tests. We are conducting serology testing within the community for SARS-CoV-2-specific antibodies through a serologic test could give insight into past COVID-19 infections within our community.

DETAILED DESCRIPTION:
Adult participants aged 18 or greater will be recruited from the greater Kingman AZ area through social media, radio, newspaper, and a press release. Participants self-selected inclusion in the study by calling into a COVID-19 hotline and will be included in the sample data following self-report of absence of covid-19 symptoms. Participants will be scheduled for testing on the weeks of 09/28/2020 and 10/05/2020. Upon recruitment, participants will be asked to complete a demographic and behavioral survey, assessing socioeconomic status, interpersonal interactions, personal protective measures, and COVID-19 symptomology in the preceding two months. Two months after initial testing, all negative SARS-CoV-2-specific antibodies participants will be contacted for repeat testing and surveying.

SARS-CoV-2-specific antibodies will be tested using a lateral flow immunoassay with the VITROS Anti-SARS-CoV-2 IgG test (Ortho-Clinical Diagnostics, Inc.) under the Emergency Use Authorization (EUA) from the Food and Drug Administration (FDA). The diagnostic sensitivity of the immunoassay was 87.5% and specificity was 100%. The positive and negative predictive value with a prevalence of 5% in the community was 100% and 99.3% respectively. All data will be de-identified and stored in a password protected file only visible to study investigators. All positive results were called back to participants by the lead author.

Data obtained was then used to estimate the population prevalence of SARS-CoV-2-specific antibodies in the Kingman, Arizona population. Unweighted and weighted proportions of positive tests were calculated to match the 2018 census on sex, race, education, and income. Confidence intervals for unweighted data will be estimated using exact binomial models and for weighted and adjusted estimates using bootstrap methods. All data was analyzed using SPSS.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18+
* Resident of Mohave County AZ

Exclusion Criteria:

* Children under 18yo
* Previous positive SARS-CoV2- Antibody Test
* Active symptoms of respiratory Illness

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: ~30,000 individuals inhabit Kingman AZ across 7,854 households, out of which 30.1% had children under the age of 18 living with them, 54.6% were married couples living together, 10.1% had a female householder with no husband present, and 30.9% were non-families. 25.5% of all households were made up of individuals, and 11.7% had someone living alone who was 65 years of age or older.
Sampling Method: Probability Sample
Enrollment: 566 (Actual)
Dates: Start 2020-09-28 (Actual); Primary Completion 2020-10-09 (Actual); Study Completion 2021-05-01 (Actual)

PRIMARY OUTCOMES:
Seroprevelence of SARS-CoV-2 Antibodies among Adults in Kingman AZ | 2-weeks
  A sample from the population of Kingman AZ will be used to determine the epidemiology of COVID-19 spread throughout Kingman AZ.

SECONDARY OUTCOMES:
Retention of SARS-CoV-2 Antibodies among Adults in Kingman AZ | 2-weeks
  Participants will have a second antibody diagnostic test 2 months following initial enrollment. The concordance between positive tests will then be used to determine the longevity of SARS-CoV-2 antibodies in our community.

CONTACTS AND LOCATIONS:
Overall Officials: Anthony J Santarelli, PhD, Study Director — Kingman Healthcare Inc.
Locations (1):
- Kingman Regional Medical Center, Kingman, Arizona, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Paul R, Arif AA, Adeyemi O, Ghosh S, Han D. Progression of COVID-19 From Urban to Rural Areas in the United States: A Spatiotemporal Analysis of Prevalence Rates. J Rural Health. 2020 Sep;36(4):591-601. doi: 10.1111/jrh.12486. Epub 2020 Jun 30. PMID 32602983
- [Background] Peters DJ. Community Susceptibility and Resiliency to COVID-19 Across the Rural-Urban Continuum in the United States. J Rural Health. 2020 Jun;36(3):446-456. doi: 10.1111/jrh.12477. Epub 2020 Jun 16. PMID 32543751
- [Derived] Santarelli A, Lalitsasivimol D, Bartholomew N, Reid S, Reid J, Lyon C, Wells J, Ashurst J. The seroprevalence of SARS-CoV-2 in a rural southwest community. J Osteopath Med. 2021 Feb 1;121(2):199-210. doi: 10.1515/jom-2020-0287. PMID 33567087